CLINICAL TRIAL: NCT00310115
Title: Smoking Relapse Prevention Among Postpartum Women
Brief Title: Motivational Counseling in Preventing Smoking Relapse After Pregnancy in Pregnant Women Who Quit Smoking During Pregnancy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BS01-178; R01CA089350 (NIH); P30CA016672 (NIH); MDA-BS01-178 (Other: UT MD Anderson Cancer Center); CDR0000466327 (Registry Identifier: NCI PDQ); NCI-2010-01136 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Bladder Cancer; Cervical Cancer; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Leukemia; Liver Cancer; Lung Cancer; Pancreatic Cancer; Tobacco Use Disorder
Keywords: non-small cell lung cancer; small cell lung cancer; bladder cancer; cervical cancer; esophageal cancer; gastric cancer; renal cell carcinoma; adult primary liver cancer; pancreatic cancer; hypopharyngeal cancer; lip and oral cavity cancer; laryngeal cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; adult acute myeloid leukemia; tobacco use disorder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Tobacco Use Disorder; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Hypopharyngeal Neoplasms; Mouth Neoplasms; Laryngeal Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Leukemia, Myeloid, Acute | interventions — Counseling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Smoking Prevention Usual Care: Arm I (usual care): Self-help materials and brief relapse prevention advice based on Treating Tobacco Use and Dependence Clinical Practice Guideline.
  Interventions: Behavioral: Smoking Prevention Usual Care
- MRP: Arm II (motivational relapse prevention [MRP]): Same intervention as usual care, plus 30 minutes telephone counseling at 34 & 36 weeks gestation then at 2, 4, 7, & 16 weeks postpartum.
  Interventions: Behavioral: Smoking Prevention Usual Care; Behavioral: Counseling Intervention
- Enhanced MRP +: Arm III (enhanced MRP [MRP+]): Same intervention as usual care and telephone counseling as MRP, plus 1 hour in-person counseling at 30-33 weeks gestation & 8 weeks postpartum.
  Interventions: Behavioral: Smoking Prevention Usual Care; Behavioral: Counseling Intervention

INTERVENTIONS:
Behavioral: Smoking Prevention Usual Care — Usual care of self-help materials and advice for staying cigarette free
Behavioral: Counseling Intervention — 6 x 30 minute counseling sessions over the telephone
  Groups: Enhanced MRP +; MRP
Behavioral: Counseling Intervention — 2 in-person counseling sessions
  Groups: Enhanced MRP +

SUMMARY:
RATIONALE: Motivational counseling may help prevent pregnant women from smoking again after pregnancy.

PURPOSE: This randomized clinical trial is studying three different types of counseling to see how well they work in preventing smoking relapse after pregnancy in pregnant women who quit smoking during pregnancy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop and evaluate 2 "Motivational Relapse Prevention" (MRP) treatments of varying intensity for reducing postpartum smoking relapse among pregnant women who quit smoking during pregnancy.
* Assess MRP and Enhanced MRP (MRP+) effects on treatment mechanisms and the role of those mechanisms in mediating MRP and MRP+ effects on abstinence.
* Assess the cost-effectiveness of both the MRP and MRP+ treatments relative to each other and to usual care for reducing postpartum smoking relapse.

OUTLINE: This is a randomized study. Participants are randomized to 1 of 3 intervention arms.

* Arm I (usual care [UC]): Participants receive self-help materials and brief relapse prevention advice based on the Treating Tobacco Use and Dependence Clinical Practice Guideline.
* Arm II (motivational relapse prevention [MRP]): Participants receive the same intervention as in arm I. Participants also undergo telephone counseling over 30 minutes at 34 and 36 weeks gestation and then at 2, 4, 7, and 16 weeks postpartum.
* Arm III (enhanced MRP [MRP+]): Participants receive the same intervention as in arm I and telephone counseling as in arm II. Participants also undergo in-person counseling over 1 hour at 30-33 weeks gestation and then at 8 weeks postpartum.

Participants in all arms complete questionnaires at baseline, at 30-33 weeks gestation, and then at 8 and 26 weeks postpartum.

Participants are followed at 8 and 26 weeks postpartum.

PROJECTED ACCRUAL: A total of 450 participants will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older
2. former smoker who quit during pregnancy as assessed via self-report
3. smoked an average of greater than or equal to 1 cigarette per day during the year prior to the current pregnancy
4. gestational age < 33 weeks and ability to attend an in-person visit at University of Texas MD Anderson Cancer Center (UTMDACC) between 30-33 weeks of gestational age
5. can speak, read and write in English.
6. must have a functioning home or personal cell phone

Exclusion Criteria:

1) high-risk pregnancy or known negative birth outcome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, 18 years of age or older, who quit smoking while pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2002-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Smoking Abstinence | 26 weeks
  Smoking abstinence as measured by the Society for Research on Nicotine and Tobacco Smoking Status Measure at 26 weeks following study treatment

SECONDARY OUTCOMES:
Number of Cigarettes Smoked Daily | 26 weeks following study treatment
  Cigarettes smoked per day at 26 weeks following study treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, PhD, BS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org